CLINICAL TRIAL: NCT07278791
Title: A Survey-Based Study on Differences in Recovery Periods of Upper Extremity Injuries Among Indoor Climbers According to Treatment Methods
Brief Title: Survey-Based Study on Recovery Period Differences in Upper Extremity Injuries Among Indoor Climbers by Treatment Method
Status: Not yet recruiting | Type: Observational
Sponsor: Sahmyook University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-06-034-002
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Upper Extremity Injury
Keywords: Indoor Climbing; Bouldering; Physical Therapy; Self-Treatment; Rehabilitation; Injury Recovery; Upper Limb; Sports Injury
MeSH Terms: conditions — Arm Injuries; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Self-Treatment Group: Participants who treated their upper extremity injury through self-managed care such as rest, cold/heat therapy, taping, or over-the-counter medication.
- Physical Therapy Group: Participants who received professional non-surgical physical therapy, including manual therapy, therapeutic exercise, or extracorporeal shockwave therapy.
- Injection Therapy Group: Participants who received non-surgical injection treatments such as prolotherapy, PRP, or steroid injections for upper extremity injury.
- Surgery/Rehabilitation Group: Participants who underwent surgical or invasive procedures followed by rehabilitation or exercise-based recovery programs.

SUMMARY:
This study aims to investigate the differences in recovery periods of upper extremity injuries among indoor climbers according to their treatment methods.

The research focuses on comparing the recovery duration, specifically the time to return to climbing, between those who received professional physical therapy and those who relied on self-treatment or other conservative management.

Additionally, this survey-based observational study seeks to explore how individual and training-related factors - such as warm-up duration, climbing frequency, and years of experience - affect the occurrence and recurrence of upper extremity injuries.

Participants will complete an online questionnaire consisting of demographic data, climbing habits, injury characteristics, treatment methods, and recovery outcomes.

The data will be collected anonymously and analyzed to determine whether the type of treatment correlates with faster recovery or reduced reinjury risk.

The findings are expected to provide foundational evidence for developing effective rehabilitation and injury-prevention strategies for indoor climbers, and to guide clinicians and trainers in selecting appropriate treatment approaches for upper extremity injuries.

DETAILED DESCRIPTION:
This cross-sectional survey will recruit indoor climbers aged 18-50 who have experienced upper extremity injuries within the past 12 months.

The questionnaire includes sections on injury site and type (e.g., finger, wrist, elbow, shoulder; tendonitis, ligament injury, or muscle tear), treatment method (self-care, physical therapy, injection, surgery, or rehabilitation exercise), treatment duration, and perceived recovery status.

Statistical analysis will be performed to compare mean recovery periods among treatment groups and to examine correlations with demographic and behavioral factors.

The study was approved by the Institutional Review Board of Sahmyook University (IRB No. 2025-06-034-002).

Results from this research may contribute to improved understanding of injury management and evidence-based rehabilitation for indoor climbers.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years.
* Individuals who have participated in indoor climbing within the past 12 months.
* Individuals who have experienced an upper extremity injury (e.g., finger, wrist, elbow, shoulder; tendonitis, ligament injury, muscle tear) during indoor climbing within the past 12 months.
* Individuals who received any form of treatment (self-care, physical therapy, injection, surgery, rehabilitation exercise) for the injury.
* Individuals who can provide informed consent and complete an online questionnaire.

Exclusion Criteria:

* Individuals who underwent major orthopedic surgery or fracture-related surgery unrelated to climbing.
* Individuals who required hospitalization or long-term inpatient treatment (>3 months) due to severe musculoskeletal conditions.
* Individuals currently receiving ongoing treatment for the same injury.
* Individuals with neurological, systemic, or medical conditions that significantly affect musculoskeletal recovery.
* Climbing coaches, professional climbers, or clinicians providing treatment (to avoid expert bias).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will include indoor climbers aged 18 to 50 who experienced an upper extremity injury related to climbing within the past 12 months and received any form of treatment. Participants will be recruited from climbing communities, gyms, and online platforms. Only non-professional climbers will be included to ensure generalizability to the general indoor climbing population.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mean Recovery Duration (Weeks) According to Treatment Type | 12 months (retrospective survey)
  The average number of weeks required for indoor climbers to achieve full recovery and return to climbing after upper extremity injury, compared across treatment types (self-care, physical therapy, injection, surgery/rehabilitation).

SECONDARY OUTCOMES:
Reinjury Rate Within 12 Months | 12 months
  Proportion of indoor climbers who experienced a recurrent upper-extremity injury in the same anatomical region within the past 12 months.
Pain Resolution Duration (Weeks) | 12 months (retrospective survey)
  Number of weeks required for complete pain resolution after upper-extremity injury, based on participant recall.
Return-to-Climbing Criteria (Self-Reported) | 12 months
  Self-reported criteria participants used to determine readiness to resume climbing after upper-extremity injury (e.g., full pain resolution, daily activity tolerance, strength recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Changyong Choi, PT, MPT Candidate, Principal Investigator — Sahmyook University; Seungwon Lee, PhD, PT, Study Chair — Sahmyook University

IPD SHARING:
Plan to Share IPD: No
This study does not collect individual participant data (IPD) such as raw clinical data or identifiable records. All survey responses are anonymized, aggregated, and analyzed at the group level. Therefore, there is no IPD available to share.

REFERENCES:
- [Background] Schoffl V, Popp D, Kupper T, Schoffl I. Injury trends in rock climbers: evaluation of a case series of 911 injuries between 2009 and 2012. Wilderness Environ Med. 2015 Mar;26(1):62-7. doi: 10.1016/j.wem.2014.08.013. PMID 25712297